CLINICAL TRIAL: NCT06364111
Title: Comparative Study on the Efficacy of Disposable Gastrointestinal Vibrating Capsule (Vibrabot Capsule) and Polyethylene Glycol for Chronic Functional Constipation
Brief Title: Comparative Study on the Efficacy of Vibrabot Capsule and Polyethylene Glycol for Chronic Functional Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vibrabot Capsule
Record Dates: First submitted 2023-12-12; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2023-12

CONDITIONS: Chronic Functional Constipation
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trial group 1 (Experimental): Subjects in Trial Group 1 received polyethylene glycol combined with Vibrabot capsules for 2 weeks and then Vibrabot capsules for 4 weeks.
  Interventions: Device: Vibrabot capsule
- Trial group 2 (Experimental): Subjects in Trial Group 2 received Vibrabot capsules for 12 consecutive weeks.
  Interventions: Device: Vibrabot capsule
- Control group (Experimental): subjects in the control group received polyethylene glycol for 6 weeks.
  Interventions: Drug: polyethylene glycol

INTERVENTIONS:
Device: Vibrabot capsule — Subjects in Trial Group 1 received polyethylene glycol combined with Vibrabot capsules for 2 weeks and then Vibrabot capsules for 4 weeks; Subjects in Trial Group 2 received Vibrabot capsules for 12 consecutive weeks.
  Arms: Trial group 1; Trial group 2
Drug: polyethylene glycol — Subjects in the control group received polyethylene glycol for 6 weeks
  Arms: Control group

SUMMARY:
This is a single-center trial that enrolls 20 18 to 85-year-old patients with moderate to severe FC to study the efficacy of Vibrabot capsule (dosage: 5 capsules/week) and polyethylene glycol, as well as the mechanism of action of the Vibrabot capsule.

DETAILED DESCRIPTION:
This study is a prospective, parallel controlled clinical trial. Subjects are considered eligible for this study if they meet the inclusion criteria and do not meet any of the exclusion criteria. They must sign an Ethics Committee (EC)-approved Informed Consent Form (ICF) and be randomly assigned to trial group 1, trial group 2 and control group for the respective treatment.

Subjects in Trial Group 1 received polyethylene glycol combined with Vibrabot capsules for 2 weeks and then Vibrabot capsules for 4 weeks; Subjects in Trial Group 2 received Vibrabot capsules for 12 consecutive weeks; Subjects in the control group received polyethylene glycol for 6 weeks, and subjects with poor efficacy could voluntarily choose to continue to receive Vibrabot capsules for 6 weeks. During the treatment period, the dosage of Vibrabot capsule is 1 capsule/time, 5 times/week, and that of polyethylene glycol is 10g/time, twice/day. The subjects who receive Vibrabot capsules will undergo a colonic transit study, a radionuclide imaging-based gastrointestinal transit assessment, an anorectal manometry, a neurotransmitter test, and a fecal flora test before and after the treatment. After completion of treatment, subjects in each group entered a follow-up period, which was observed until the patient regained symptoms of constipation, i.e., when laxatives or other bowel-promoting treatments were used. If the subject never recovered from constipation, a minimum of 8 weeks of questionnaire completion was required, depending on the patient's compliance status. During the study period, the subjects are required to keep an e-diary recording daily bowel movements (BMs), medication intake, and discomforts, and complete the Patient Assessment of Constipation-Symptoms (PAC-SYM) and the Patient Assessment of Constipation Quality of Life (PAC-QOL) questionnaires every two weeks.

This study consists of a screening/baseline period, a treatment period and a follow-up period. During the study, subjects are required not to change their diet and lifestyle. The washout or follow-up period will end once the subject uses rescue medication. If subjects have no BM for three or more consecutive days, they are permitted to take bisacodyl as rescue medication. If they cannot tolerate bisacodyl, an enema may be used instead. They should avoid antibiotics, probiotics, prebiotics, and proton pump inhibitors throughout their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

1. People with moderate to severe functional constipation according to Rome IV criteria.
2. People who agree to use appropriate medical methods of contraception from the time they sign the ICF until the end of the treatment period (excluding women in a medical sterilization status).
3. People who had a colonoscopy within three years before screening and negative results, or their colonoscopy results are judged by the investigator as mild anomalies, but the cause of their constipation cannot be explained. If the colonoscopy report is unavailable, the study physician will determine if a colonoscopy is needed. If the subjects undergo a colonoscopy after signing the ICF, they will not enter the treatment period until their BMs return to the baseline level.
4. People had colonic polyps and a polypectomy (except for endoscopic submucosal dissection (ESD)): Those with a polyp ≤1 cm can be enrolled one month after the polypectomy; Those with a polyp >1 cm can be enrolled three months after the polypectomy.
5. People who consent to participate in this trial and can communicate with the investigator and can understand and comply with the relevant procedures and requirements during the study (including completing study questionnaires on time, being treated and visited as scheduled, and undergoing relevant examinations), and voluntarily sign the ICF.

Exclusion Criteria:

1. People who are not eligible for surgery or refuse to undergo any abdominal surgery.
2. People with known or suspected gastrointestinal obstruction, stenosis, diverticulum, bleeding, malformation, and fistula.
3. People allergic to polymeric materials.
4. People implanted with cardiac pacemakers and using gastrointestinal pacemakers.
5. People with abdominal aortic aneurysms, gastrointestinal vascular lesions, ulcers, and lesions with bleeding tendencies.
6. People with dysphagia.
7. Pregnant women or women with pregnancy plans in the next year.
8. People with severe depression and anxiety and severe acute gastrointestinal lesions.
9. People who had gastrointestinal surgery or a history of surgery that changed the structure of the gastrointestinal tract (except for appendectomy) or people who underwent gastrointestinal ESD in the past three months.
10. People with severe hemorrhoids (patients with grade III-IV hemorrhoids according to the Clinical Practice Guidelines for the Management of Hemorrhoids of the American Society of Colon and Rectal Surgeons).
11. People who plan to undergo MRI in the near future.
12. People with other conditions, so the investigator considers them not eligible for this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-06-14 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
The proportions of responders to the three therapies during the treatment period. | 18 months
  Responders are the subjects with an average increase of ≥1 complete spontaneous bowel movements (CSBMs) per week during the treatment period compared to the baseline period.

SECONDARY OUTCOMES:
Evaluation of intestinal motility | 18 months
  Comparison of colonic transit time (h) before and after treatment with Vibrabot capsules.
Assessment of neurotransmitters in peripheral blood | 18 months
  Changes in peripheral blood levels (ng/ml) of five neurotransmitters, NO, VIP, 5-HT, SP, and GABA, before and after treatment with Vibrabot capsules.
Assessment of changes in intestinal flora | 18 months
  Assessment of changes in intestinal flora.
Evaluation of the treatment cycle of Vibrabot Capsules | 18 months
  Evaluate the percentage of responders to 6 weeks of treatment versus 12 weeks of treatment with Vibrabot capsules.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Jiang, Professor, Principal Investigator — Beijing Tsinghua Changung Hospital
Locations (1):
- XuanJiang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No